CLINICAL TRIAL: NCT04867590
Title: A Controlled, Randomised Multicenter Study Comparing the Effectiveness of EndoRotor (New Treatment Technique) Versus Radiofrequency (Reference Technique) in Treating Barrett's Esophagus Complicated by Dysplasia
Brief Title: A Study Comparing the Effectiveness of EndoRotor Versus Radiofrequency in Treating Barrett's Esophagus
Acronym: ENDOBARRETT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00975-34
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Barrett Esophagus; Dysplasia
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EndoRotor (Experimental): The ENDOROTOR is a new system for the resection of superficial lesions within the digestive tract and composed of a reusable generator, a single-use probe and additional accessories.
  The device is used in the resection of mucosa in the digestive tract: flat or slightly raised lesions in the digestive mucosa, or treatment of the lateral margins following a resection carried out using another technique.
  Resected tissue is aspirated away through a rotating catheter: the cutting and removal of tissue as well as the collection of specimens are combined into one act.
  Interventions: Device: Endorotor
- Radiofrequency (Active Comparator): Endoscopic treatment using the HALO® 360 or 90 system is a thermal ablation system for superficial mucosa. First and foremost, the examination includes an endoscopy to locate the upper limits of the BE and its distribution, so as to choose the most appropriate type of probe. An initial debridement of the mucosal deposits is carried out by application of acetylcysteine in spray form with a spray catheter on the entire mucosal surface to be treated and then rinsed with water after a minute of application time.
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Device: Endorotor — The treatment itself is preceded by a sub-mucosa saline and adrenalin solution injection administered by an endoscopic sclerotherapy needle lifting the submucosa and thus reducing the risk of perforation and hemorrhage.
  The interventional tool is then applied tangentially to be brought into contact with the lifted mucosa, visual monitored by endoscope. The aspiration and sectioning system is activated by use of a pedal and a generator specially made for the system, used in every procedure. The entire surface area of the targeted mucosa must be covered by the probe. The residual tissue is then removed via the aspiration system and caught by a filter. The specimens are then easily retrievable at the end of the procedure and can be stored in formalin fixing solution for histological analysis.
  Arms: EndoRotor
Device: Radiofrequency — Endoscopic treatment using the HALO® 360 or 90 system is a thermal method for destroying the superficial mucosa. An initial debridement of the mucosal deposits is carried out by application of acetylcysteine in spray form with a spray catheter on the entire mucosal surface to be treated and then rinsed with water after a minute of application time.
  For circumferential BEs, a single-use 360 Express® probe is used to make it possible to size the diameter of the esophagus and the treatment used. The length of the treatment area is 5 cm and several points of impact can be achieved by overlapping the catheter at two consecutive heights, with the zone spanned measuring one centimeter, in order to cover the entire pathological area requiring treatment.
  For non-circumferential lesions a "palette" applicator is used in a variety of sizes, and in this context no sizing of the esophagus is required.
  Arms: Radiofrequency

SUMMARY:
Barrett Esophagus is a common pathology, with an estimated prevalence of 1.6% at risk of progression to precancerous mucosa (low to high grade dysplasia). The incidence of adenocarcinoma on BE is 0.5% per year. In the event of dysplasia or cancer in situ, it is currently recommended at international and particularly European level to eradicate BE. The treatment techniques used to date carry out thermal destruction of the BE, in particular by radiofrequency. Eradication of dysplasia is achieved in 81% to 100% and disappearance of BE in 73% to 87% of cases. It requires an average of 3 destruction sessions. RF does not allow histological analysis after destruction of BE, but the risk of progression to neoplasia is estimated at 7.8/1000 persons per year. This risk could be due to the presence of glands buried in the esophageal mucosa. Indeed, these glands are not destroyed by thermal ablation methods, and remain invisible during endoscopic controls.

A new treatment technique using the Endorotor® system allows mechanical resection of the entire mucosa in one session of treatment. In addition, the cost of these thermal destruction techniques currently limits their wider diffusion. It is therefore legitimate to propose a less expensive and probably more effective alternative technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting Barrett's esophagus of a size between 2 cm and 6 cm in the height of the longest tonguea with low to high grade dysplasia that is histologically proven or with a superficial non-invasive adenocarcinoma that has been resected a The total height of the BE is evaluated according to the Prague classification, with the height of the circumferential segment between 0 cm (non-circumferential segment) and 6 cm (segment shaped like a full sleeve for 6 cm), referred to as C0 to C6, and the height of the longest tongue between 2 cm and 6 cm (M2- M6).
* Patients must have signed the consent form in order to participate in the study
* Patients are pre-included (signature of consent) before the histological confirmation of dysplasiab and/or superficial non-invasive adenocarcinoma that allows the patient to be included in the study.

Exclusion Criteria:

* Individuals over 85 years old
* Women who are pregnant, breastfeeding or in labour
* Individuals in detention through judicial or administrative decision
* Individuals who are the subject of psychiatric treatment under duress
* Individuals who are subjects of legal protection measures
* Individuals who are in no state to give their consent
* Individuals who do not understand French or do not know how to read
* Individuals who are not part of a social security program or benefit from such a scheme
* Those with active peptic and/or radiation-induced or complicated esophagitis at the time of treatment
* Presence of a visible lesion that is suspected to be esophageal cancer confirmed by biopsies
* Anterior resection of invasive adenocarcinoma using endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) with invasion of the lateral and/or deep margin, adenocarcinoma of poorly differentiated characteristics or sub-mucosal invasion > 500µm (pT1b)
* All preliminary ablation treatments or dilation for esophageal stenosis
* Significant esophageal stenosis: cannot be passed with a standard gastroscope
* Presence of esophageal varices or portal hypertension
* Anticoagulant treatment that cannot be stopped before the intervention (excluding 100 mg maximum per day of aspirin in single-drug treatment) or any haemostasis problems that cannot be corrected
* Having a contraindication regarding anaesthesia
* Patients incapable of taking proton pump inhibitors (PPIs) orally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The rate of full eradication of Barrett esophagus (metaplasia), which is defined by the absence of residual Barrett esophagus in the check-up endocopy after 3 months | 3 months after the endoscopic treatment
  To evaluate, 3 months after the first endoscopic treatment, the effectiveness of Endorotor treatment versus Radiofrequency in the elimination of Barrett esophagus complicated with dysplasia or adenocarcinoma.

SECONDARY OUTCOMES:
Effectiveness assessment defined by the absence of dysplasia on all systematic esophageal biopsies confirmed by a double anatomical pathological reading on site, with centralised re-reading in the event of disagreement | 3 months after the initial endoscopic treatment
  To compare the effectiveness of endoscopic Endorotor treatment versus Radiofrequency esophageal treatment on eradication of dysplasia 3 months after the initial endoscopic treatment
Effectiveness assessment defined by the absence of dysplasia on all systematic oesophageal biopsies confirmed by a double anatomical pathological reading on site, with centralised re-reading in the event of disagreement | 12 months after the initial treatment
  To compare the effectiveness of endoscopic Endorotor treatment versus Radiofrequency esophageal treatment on eradication of dysplasia 12 months after the initial treatment
Effectiveness assessment defined by the area regression of Barrett esophagus between the pre-treatment evaluation and the follow-up at 3 months is evaluated using a visual endoscopic scale of the area Barrett esophagus regression | 3 months after the initial endoscopic treatment
  To compare the effectiveness of endoscopic Endorotor treatment versus Radiofrequency esophageal treatment on the area of Barrett esophagus regression 3 months after the initial treatment
Effectiveness assessment defined by the area regression of Barrett esophagus between the pre-treatment evaluation and the follow-up at 12 months is evaluated using a visual endoscopic scale of the area Barrett esophagus regression | 12 months after the initial treatment
  To compare the effectiveness of endoscopic Endorotor treatment versus Radiofrequency esophageal treatment on the area of Barrett esophagus regression 12 months after the initial treatment
Effectiveness assessment defined by the rate of eradicating Barrett esophagus 12 months after the initial endoscopic treatment which is confirmed by the absence of Barrett esophagus lesions on biopsies | 12 months after the first treatment
  To compare the effectiveness of endoscopic Endorotor treatment versus Radiofrequency esophageal treatment on eradication of Barrett esophagus 12 months after the first treatment
Effectiveness assessment defined by the number of additional treatment sessions carried out using radiofrequency to achieve complete eradication of Barrett esophagus at 12 months, after initial endoscopic treatment | 12 months after the initial treatment
  To compare the effectiveness of endoscopic Endorotor treatment versus Radiofrequency esophageal treatment to determine the number of additional sessions carried out to achieve complete eradication at 12 months after the initial treatment
Safety assessment defined by the discomfort score is recorded in a log over as well as dysphagia score and pain evaluation in first 30 days following the initial procedure and during the clinical evaluating | 3 months after the initial endoscopic treatment
  After 3 months, evaluating the safety of endoscopic treatment with Endorotor, compared to the reference treatment with esophageal radiofrequency to evaluating clinical tolerance
Safety assessment defined by the serious adverse events after treatment and then at day 2, day 15, day 30 and 3 months after the initial endoscopic treatment are classed in four levels of severity based on the level of hospitalization, in accordance with | 3 months after the initial treatment
  After 3 months, evaluating the safety of endoscopic treatment with Endorotor, compared to the reference treatment with esophageal radiofrequency to register the rate of serious adverse events
Safety assessment defined by esophageal stenosis that cannot be passed by a standard gastroscope of 10 mm in diameter. | 3 months after the initial treatment
  After 3 months, evaluating the safety of endoscopic treatment with Endorotor, compared to the reference treatment with esophageal radiofrequency to evaluate the rate of esophageal stenosis
Evaluating the benefit of anatomo pathological analysis of resected tissue after treatment using ENDOROTOR defined by the quality of the anatomical pathological analysis for the samples taken during treatment is determined through a centralised readin | 12 months after the first treatment
  Evaluate benefits of histological information obtained with Endorotor to evaluate the quality of anatomical pathology analysis of resected samples using Endorotor
Evaluating the benefit of anatomo pathological analysis of resected tissue after treatment using ENDOROTOR defined by the percentage of patients for whom the analyses of resected tissue enable the discovery of a dysplasia or adenocarcinoma | 12 months after the first treatment
  Determine percentage of patients for whom the analysis of resected tissue will enable the discovery of a dysplasia or adenocarcinoma, ignored on the first biopsies
Evaluating the benefit of anatomo pathological analysis of resected tissue after treatment using ENDOROTOR defined by the percentage of patients for whom the analyses of resected tissue enable a change in the follow-up plan | 12 months after the first treatment
  Determine percentage of patients for whom the analysis of resected tissue will enable a change in their follow up
Evaluating the efficiency defined by the incremental cost-utility ratio | 12 months after the first treatment
  To assess and compare the efficiency of endoscopic EndoRotor treatment against radiofrequency treatment in the elimination of Barrett's eosophagus in term of cost per Quality Adjusted Life Years gained
Evaluating the efficiency defined by the incremental cost-effectiveness ratio | 12 months after the first treatment
  To assess and compare the efficiency of endoscopic EndoRotor treatment against radiofrequency treatment in the elimination of Barrett's eosophagus in term of cost per rate of eradicating barrett's eosophagus
Build a model to predict incomplete response for eradication of Barrett's eosophagus on the basis of each independent predictor coefficient in the multivariate regression logistic model | 12 months
  Build a predictive model of incomplete response to eradication of Barrett's eosophagus

CONTACTS AND LOCATIONS:
Overall Officials: Elodie CESBRON-METIVIER, Ph.D., Principal Investigator — UH Angers
Locations (12):
- France (12):
  - University Hospital of Brest, Brest
  - University Hospital of Tours, Chambray-lès-Tours
  - University Hospital of Lille, Lille
  - University Hospital of Limoges, Limoges
  - Edouard Herriot Hospital, Lyon
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - Cochin Hospital, Paris
  - Georges Pompidou European Hospital, Paris
  - University Hospital of Bordeaux, Pessac
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided